CLINICAL TRIAL: NCT02338947
Title: A Multicenter, Prospective, Randomized, Clinical Trial Comparing Off-pump Versus On-pump Coronary Artery Bypass Grafting in Frail Patients
Brief Title: Off-pump Versus On-pump Coronary Artery Bypass Grafting in Frail Patients
Acronym: FRAGILE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Beneficência Portuguesa de São Paulo (Other); Instituto Nacional de Cardiologia de Laranjeiras (Other); Clinical Hospital Samuel Libânio of Pouso Alegre (Unknown); Hospital do Coração de Messejana Dr. Carlos Alberto Studart (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USaoPauloGH1000; Sao Paulo Research Foundation (Other Grant/Funding Number: 2015/23972-3)
Record Dates: First submitted 2014-08-29; First posted 2015-01-15 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-01

CONDITIONS: Frail Elderly; Coronary Artery Disease
Keywords: Frail elderly; Coronary artery bypass surgery; Off-pump; On-pump; Randomized controlled trial
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly assigned to off-pump CABG or on-pump CABG procedure.
Who Masked: Participant, Outcomes Assessor
Masking Description: Treatment assignments will be performed in a blinded manner according to a blocked randomization scheme with a block size of ten, stratified according to the participating center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Off-pump coronary-artery bypass grafting - OPCAB (Active Comparator): Pre-frail and frail patients will be randomly assigned to OPCAB after the evaluation of the target vessels by an internet-based, password protected database program. The surgery will be performed as described in the "intervention" section and the patients will be followed up for two years.
  Interventions: Other: Off-pump coronary-artery bypass grafting
- On-pump coronary-artery bypass grafting - CABG (Active Comparator): Pre-frail and frail patients will be randomly assigned to CABG after the evaluation of the target vessels by an internet-based, password protected database program. The surgery will be performed as described in the "intervention" section and the patients will be followed up for two years.
  Interventions: Other: On-pump coronary-artery bypass grafting

INTERVENTIONS:
Other: Off-pump coronary-artery bypass grafting — Surgical access to the heart will be gained through a median sternotomy in all of the patients. In order to reduce the risk of bleeding and transfusions, an absorbable hemostat will be used in the sternal bone marrow. An automatic autotransfusion system will be used to recovery of red blood cells in all patients. Off-pump surgery will be performed with the use of heart stabilizers. Patients will be heparinized with 250 IU/kg intravenously to achieve activated clotting time >200s. The proximal anastomosis will be performed according to our guidelines. The distal anastomosis will be constructed with the help of mechanical stabilizers and cardiac positioner. Intracoronary shunts will be used routinely.
  Other Names: OPCAB
  Arms: Off-pump coronary-artery bypass grafting - OPCAB
Other: On-pump coronary-artery bypass grafting — Surgical access to the heart will be gained through a median sternotomy in all of the patients. On-pump surgery will be performed in normothermia, with the use of aortic cross-clamping and cold cardioplegic arrest. Patients will be heparinized with 500 IU/kg to achieve an activated clotting time >480 s. Heparin will be neutralized with 1:1 protamine sulfate. The automatic autotransfusion system will be used just in massive blood loss to recovery the red blood cells. Surgical techniques will be performed according to our guidelines.
  Other Names: CABG
  Arms: On-pump coronary-artery bypass grafting - CABG

SUMMARY:
Frailty is defined as a geriatric syndrome of impaired resiliency to stressors (such as cardiac surgery) that has been delineated recently in the cardiovascular literature. One of the most controversial areas of cardiac surgery has been whether off-pump coronary artery bypass grafting (OPCAB) surgery is superior to conventional on-pump coronary artery bypass grafting (CABG) surgery. There is an ongoing debate about the benefits and disadvantages of OPCAB surgery and we believe that this remains an important technique for the improvement of coronary surgery. The benefits of CABG surgery in frail patients are still undetermined. The aim of this study is to clarify the potential benefit of OPCAB surgery in pre-frail and frail patients by comparing off-pump versus on-pump CABG in these patients.

DETAILED DESCRIPTION:
The FRAGILE protocol is a national multicenter randomized controlled trial (RCT), conducted in 6 Brazilian institutions. The study is already approved by a certified ethics committee. Funding is provided by a grant from São Paulo Research Foundation (FAPESP), which otherwise will not have any role in the conduct of the study nor in the analysis nor in the reporting of data. A confidentiality agreement regarding data use and the data safety will be monitored by an independent monitoring board. All the authors will provide revisions and comments and be testifying for the accuracy and completeness of the report, as well as for the fidelity of the report to the study protocol.

ELIGIBILITY:
Inclusion criteria:

- Participants aged ≥60 years with the indication of myocardial revascularization with ≥2 criteria of frailty by Fried Frailty Criteria, and suitable to undergo either Off-pump or On-pump CABG.

Exclusion criteria:

- Patients with the indication of angioplasty or another procedure in addition to CABG; patients who underwent an emergency operation (within 24 hours after hospital admission); patients who underwent previous cardiac surgery, even with other approaches than median sternotomy; patients who do not have free, prior and informed consent to participate in this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events after OPCAB and CABG in pre-frail and frail patients | From the date of surgery until 30 days postoperatively, assessed up to 30 days
  This composite outcome comprises: all cause death, acute myocardial infarction, stroke, renal failure, acute respiratory distress syndrome and bleeding reoperation

SECONDARY OUTCOMES:
Operative time | From the start of anesthesia induction to the end of the surgical procedure
  Operative time in minutes
Mechanical ventilation time | From the initiation of mechanical ventilation in the operating room or ICU to the time of successful extubation
  Mechanical ventilation time in hours
Hyperdynamic shock | From the date of surgery until 30 days postoperatively, assessed up to 30 days
  A cluster of symptoms that signals the onset of septic shock, often including a shaking chill, rapid rise in temperature, flushing of the skin, galloping pulse, and alternating rise and fall of the blood pressure
New onset of atrial fibrillation | From the date of surgery until 30 days postoperatively, assessed up to 30 days
  12-lead electrocardiography (ECG) to confirm the diagnosis of new onset atrial fibrillation.
Need for pacing >24 hours | From the date of surgery until 30 days postoperatively, assessed up to 30 days
  Patient who requires pacing >24 hours
Renal replacement therapy | From the date of surgery until 30 days postoperatively, assessed up to 30 days
  Any type of renal replacement therapy in a patient who does not make continued use of this
Pneumonia | From the date of surgery until 30 days postoperatively, assessed up to 30 days
  Physician or advanced practitioner documents the diagnosis in the medical record based on laboratory findings (e.g. positive sputum culture results from transtracheal fluid and/or bronchial washings) and/or radiological evidence (e.g. chest radiograph diagnostic of pulmonary infiltrates)
Length of stay in intensive care unit | From the date of surgery until ICU discharge, assessed up to 30 days
  Total time in hours in Intensive Care Unit
Length of stay in hospital | From the date of surgery until hospital discharge, assessed up to 90 days
  Total time in days in hospital
Transfusion requirement | From the date of surgery until 30 days postoperatively, assessed up to 30 days
  Number of units of red blood cells transfused
Recurrence of angina | From the date of surgery until 30 days postoperatively, assessed up to 30 days
  To analyse patient recurrence of angina according to the Canadian Cardiovascular Society (CCS)
Rate of complete revascularization | Assessed at the end of the surgical procedure, evaluated within the intraoperative period, with an estimated duration of up to 600 minutes
  To evaluate and compare the rate of complete revascularization in each of the two strategies. Complete revascularization is defined as targeting arteries larger than 1.5 mm, with stenosis greater than 70%, and a good distal bed
Evolution of frailty status | From the date of hospital discharge until 6 months postoperatively and from the date of hospital discharge until 12 months postoperatively, assessed up to 1 year
  Frailty status will be assessed based on the Fried Frailty Criteria, which includes five components: unintentional weight loss, exhaustion, weakness (grip strength), slowness (gait speed), and low physical activity. Patients will be categorized as robust (0 criteria), pre-frail (1-2 criteria), or frail (3-5 criteria) at baseline and at follow-up. Changes in frailty status over time will be evaluated to determine progression, stability, or improvement

OTHER OUTCOMES:
Delirium | From the date of surgery until 30 days postoperatively, assessed up to 30 days
  Delirium will be assessed using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) in the ICU and the Confusion Assessment Method (CAM) in the ward. According to the CAM-ICU instrument, delirium is diagnosed when features 1 and 2 are positive, along with either feature 3 or 4. The diagnosis of delirium requires the presence of baseline mental status changes, inattention, altered level of consciousness, or disorganized thinking. Patients will be evaluated with the CAM-ICU during their stay in the Intensive Care Unit and with the CAM after being transferred to the ward, but this assessment will only be conducted at the coordinating center
Neurobehavioral outcomes after cardiac surgery | From the date of hospital discharge until 6 months postoperatively and from the date of hospital discharge until 12 months postoperatively, assessed up to 1 year
  To evaluate the global cognitive status a examination test will be performed included 30 simple questions and tasks in a number of areas (orientation in time and place, repeating and recalling list of words, arithmetic, language use and comprehension, non-verbal memory)
Quality of life after cardiac surgery | From the date of hospital discharge until 6 months postoperatively and from the date of hospital discharge until 12 months postoperatively, assessed up to 1 year
  To evaluate the quality of life by the EuroQol-registration, a five domain and a visual analogue scale (VAS). The best state they can imagine is marked by 100 and the worst state marked by 0
Cost | From the date of surgery until 12 months postoperatively, assessed up to 1 year
  The adjusted amount in US dollars of the total cost of coronary artery bypass surgery will be evaluated only at the coordinating center (InCor/HCFMUSP)
Graft patency | From the date of surgery until 12 months postoperatively, assessed up to 1 year
  Patency of grafts and coronary artery disease at 1 year of follow-up evaluated by angiotomography
Clinical and angiographic scores correlation with prognostic | From the date of surgery until 12 months postoperatively, assessed up to 1 year
  To evaluate the clinical correlation between the revascularization strategy and the usefulness of the SYNergy between percutaneous coronary intervention with TAXus and cardiac surgery score (SYNTAX score); age, creatinine and ejection fraction score (ACEF score); clinical SYNTAX score; European System for Cardiac Operative Risk Evaluation (EuroSCORE II); The Society of Thoracic Surgeon´s risk model (STS score) and Índice de Predição do INStituto do CORação (InsCor) for prognostic evaluation
Evaluation of the patency of the radial artery and saphenous vein in the left coronary system after Myocardial Revascularization Surgery in patients with frailty criteria - FRAGILE TRIAL | From the date of surgery until 12 months postoperatively, assessed up to 1 year
  Primary objective
  To evaluate the patency of the RA graft in relation to the SV graft in the left coronary system in MVR surgery in patients with frailty criteria through coronary tomography angiography and bypasses with 12 months of follow-up.
  Secondary objective To evaluate the operative morbidity and mortality of patients undergoing MVR surgery where the RA graft was used in relation to the patient who underwent VS.
  To evaluate the patency of RA and SV in relation to the degree of obstruction of the treated coronary vessels

CONTACTS AND LOCATIONS:
Overall Officials: Omar AV Mejia, MD, PhD, Study Director — InCor Heart Institute; Fábio B Jatene, MD, PhD, Study Chair — InCor Heart Institute
Locations (7):
- Emory University School of Medicine, Atlanta, Georgia, United States
- Brazil (6):
  - Hospital de Messejana, Fortaleza, Ceará
  - Hospital das Clínicas Samuel Libânio, Pouso Alegre, Minas Gerais
  - Hospital Alberto Urquiza Wanderley, João Pessoa, Paraíba
  - Instituto Nacional de Cardiologia de Laranjeiras, Rio de Janeiro, Rio de Janeiro
  - Beneficência Portuguesa de São Paulo, São Paulo, São Paulo
  - Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mejia OAV, Sa MPBO, Deininger MO, Dallan LRP, Segalote RC, Oliveira MAP, Atik FA, Santos MAD, Silva PGMBE, Milani RM, Hueb AC, Monteiro R, Lima RC, Lisboa LAF, Dallan LAO, Puskas J, Jatene FB. Off-pump versus On-pump Coronary Artery Bypass Grafting in Frail Patients: Study Protocol for the FRAGILE Multicenter Randomized Controlled Trial. Braz J Cardiovasc Surg. 2017 Sep-Oct;32(5):428-434. doi: 10.21470/1678-9741-2017-0196. PMID 29211225
- See also: São Paulo Research Foundation — http://www.fapesp.br/en
- See also: Zerbini Foundation — http://www.zerbini.org.br
- See also: Brazilian Cardiovascular Society — http://www.sbccv.org.br